CLINICAL TRIAL: NCT05191069
Title: Effects of Moringa Oleifera Mouthwash in Patients Undergoing Fixed Orthodontic Appliance Treatment: a Parallel Arm, Triple Blinded, Randomized Controlled Trial
Brief Title: Effect of Moringa Oleifera Mouthwash
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MINS/69/2020 Rabia Afreen
Record Dates: First submitted 2021-12-29; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Orthodontic Appliance Complication
Keywords: Moringa Oleifera; Moringa Mouthwash; Fixed Orthodontic Treatmnet; Moringa Mouthwash in orthodontics; Orthodontics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moringa Oleifera Mouthwash (Experimental): 15ml of Moringa Oleifera mouthwash will be given to be used twice daily for 6 months.
  Interventions: Other: Moringa Oleifera Mouthwash
- Placebo Mouthwash (Placebo Comparator): The mouthwash will have all other ingredients other than Moringa Oleifera extract. Participants will be advised to use 15ml of Placebo mouthwash twice daily for 6 months.
  Interventions: Other: Placebo Mouthwash

INTERVENTIONS:
Other: Moringa Oleifera Mouthwash — 15ml of the mouthwash to be used twice daily for 6 months
  Arms: Moringa Oleifera Mouthwash
Other: Placebo Mouthwash — 15ml of the mouthwash to be used twice daily for 6 months
  Arms: Placebo Mouthwash

SUMMARY:
Improvement of oral hygiene maintenance is very important during fixed orthodontic appliance treatment to prevent the degenerative effects. Different mouthwashes are available in market but this study is being conducted to check the effects of Moring Oleifera mouth wash against the development of Gingivitis, Periodontitis, Plaque formation, Enamel Demineralization /white spot lesion, discoloration and bacterial load in dental plaque during the fixed orthodontic treatment.

DETAILED DESCRIPTION:
With the increase in desire of improved facial and dental aesthetics among all social classes, the numbers of cases being treated with fixed orthodontic appliances are increasing. It is difficult to maintain certain standard of oral hygiene with the braces on, so the iatrogenic degenerative effects of fixed orthodontic appliances are somewhat inevitable. Along with proper brushing and flossing orthodontists advise the use of mouthwash as well in order to prevent or lessen the severity of gingivitis, periodontitis, gingival hyperplasia, demineralization, white spot lesions, discoloration of teeth etc.

Plenty of mouth washes are available in market containing varying concentration of different chemicals promising to improve the oral health and reduce inflammation. But all of them having certain side effects most common being the discoloration. The focus is being shifted to natural ingredients to gain the same or even better results with minimum to zero side effects. In quest of getting closer to Mother Nature Moringa Oleifera leaf was discovered in 1785 in Indian Subcontinent.

Moringa Oleifera is a nutraceutical and well known for its anti-inflammatory, anti-microbial, anti-cancer, anti-diabetes, anti-rheumatoid arthritis, hepatoprotective, Steroid-genesis modulators and neuroprotective functions and many other properties. Its leaves evidently contain various natural anti-inflammatory and anti-oxidant substances namely flavonoid, phenolic and carotenoid. Besides, MO leaves also rich in protein, vitamin C, vitamin A, calcium and potassium. Flavonoids may act as antioxidant by scavenging free radical and protecting the cell from oxidative stress. Recently quite a lot work has been done on flavonoids in dentistry which includes anti-bacterial/anti-cariogenic effects, reduction in plague formation, Treatment in surgical wounds, reduction in dentinal hypersensitivity, treatment of periodontitis and gingivitis because of its anti-inflammatory and anti-oxidative effects.

Previously studies have been done to check the efficacy of different herbal mouthwashes but no study has been done to check the efficacy of MO leaf extract mouth wash on the oral health of the patients having fixed orthodontic treatment

ELIGIBILITY:
Inclusion Criteria:

* Young healthy subjects undergoing orthodontic treatment.
* Patients with all permanent teeth present without any oral pathology.
* Healthy gingiva with no bleeding on probing before start of orthodontic treatment and a normal pocket depth (1-3mm) on all teeth.
* No WSLs (score = 1

Exclusion Criteria:

* History of smoking, patients suffering from any systemic illness like diabetes.
* Gingivitis or an active periodontal disease.
* Carious lesions on labial/buccal surface of teeth.
* Mentally handicapped individuals

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-12-23 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Periodontal Probing Depth | 7 months
  Changes from baseline, the probing depth scale will be used to assess the pocket depth, and is graded from 0-5, 0= no No pockets>3.5mm, no calculus/overhangs, no bleeding after probing(black band completely visible). 1=No pockets>3.5mm, no calculus/overhangs, but bleeding after probing(black band completely visible). 2= No pockets>3.5mm, but supra or subgingival calculus/overhangs(black band completely visible). 3=Probing depth 3.5-5.5mm (black band partially visible, indicating pocket of 4-5mm). 4=Probing depth> 5.5mm (black band entirely within pocket, indicating pocket of 6mm or more). 5=Furcation involvement.
Plaque Index | 7 months
  Changes from base line, quantity of plaque will be assessed using plaque index, graded from 0-4, 0=Absence of microbial plaque. 1=Thin film of microbial plaque along the free gingival margin. 2=Moderate accumulation with plaque in the sulcus. 3=Large amount of plaque in sulcus or pocket along the free gingival margin.
White spot Lesions | 7 months
  Changes from the baseline, white spot lesions will be assessed visually by grading from 1-4. 1= Normal, 2= Slight, 3= Severe, 4= Cavitation.
Modified Gingival Index | 7 months
  Changes from the baseline, gingivitis will be assessed using this index graded from0-4, 0= Normal, 1=Mild inflammation, slight change in color, little change in texture of any portion of gingival unit. 2= Mild inflammation of entire gingival unit. 3=Moderate inflammation of entire gingival unit. 4=Severe inflammation of entire gingival unit.
Discoloration of teeth | 7 months
  Changes from the baseline, discoloration will be assessed by taking photographs on every interval using the same camera at the same settings. these photographs will be assessed from by 2 panels 2 weeks apart.
Bacterial Load In Plaque | 3 months
  Changes from the baseline, Colony forming units will be measured by doing microbial analysis. Quantity of CFUs for S. mutans and P. Gingivalis will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Ulfat Bashir, Masters, Principal Investigator — Riphah International University
Locations (1):
- Islamic International Dental Hospital, Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Anezi SA, Harradine NW. Quantifying plaque during orthodontic treatment: Angle Orthod. 2012 Jul;82(4):748-53. doi: 10.2319/050111-312.1. Epub 2011 Nov 1. PMID 22044115
- [Background] Atanasova S, Kovachevska I, Nashkova S, Toneva V, Zlatanovska K, Longurova N. Side effects of orthodontic treatment. Knowledge International Journal. 2018;23(2):665-71
- [Background] Sioustis I, Martu M-A, Luchian I, Teodorescu C, Kappenberg-Nitescu D-C, Iovan A, et al. Clinical effects of orthodontic treatment on periodontal status. Review. Rom J of Medical and Dental Education. 2019;8(3):57-6
- [Background] Haas AN, Pannuti CM, Andrade AK, Escobar EC, Almeida ER, Costa FO, Cortelli JR, Cortelli SC, Rode SD, Pedrazzi V, Oppermann RV. Mouthwashes for the control of supragingival biofilm and gingivitis in orthodontic patients: evidence-based recommendations for clinicians. Braz Oral Res. 2014 Jul 11;28(spe):1-8. doi: 10.1590/1807-3107bor-2014.vol28.0021. Epub 2014 Jul 11. PMID 25055220
- [Background] Jeyakumar J, Sculean A, Eick S. Anti-biofilm Activity of Oral Health-care Products Containing Chlorhexidine Digluconate and Citrox. Oral Health Prev Dent. 2020 Oct 27;18(4):981-990. doi: 10.3290/j.ohpd.a45437. PMID 33215489
- [Background] Van Strydonck DA, Slot DE, Van der Velden U, Van der Weijden F. Effect of a chlorhexidine mouthrinse on plaque, gingival inflammation and staining in gingivitis patients: a systematic review. J Clin Periodontol. 2012 Nov;39(11):1042-55. doi: 10.1111/j.1600-051X.2012.01883.x. Epub 2012 Sep 7. PMID 22957711
- [Background] Dubey DK, Dora J, Kumar A, Gulsan RK. A multipurpose tree-Moringa oleifera. International Journal of Pharmaceutical and Chemical Sciences. 2013;2(1):415-23
- [Background] Sankari SL, Babu NA, Rani V, Priyadharsini C, Masthan KM. Flavonoids - Clinical effects and applications in dentistry: A review. J Pharm Bioallied Sci. 2014 Jul;6(Suppl 1):S26-9. doi: 10.4103/0975-7406.137256. PMID 25210379
- [Background] Panche AN, Diwan AD, Chandra SR. Flavonoids: an overview. J Nutr Sci. 2016 Dec 29;5:e47. doi: 10.1017/jns.2016.41. eCollection 2016. PMID 28620474
- [Background] Buakaew W, Sranujit RP, Noysang C, Sangouam S, Suphrom N, Thongsri Y, Potup P, Usuwanthim K. Evaluation of Mouthwash Containing Citrus hystrix DC., Moringa oleifera Lam. and Azadirachta indica A. Juss. Leaf Extracts on Dental Plaque and Gingivitis. Plants (Basel). 2021 Jun 6;10(6):1153. doi: 10.3390/plants10061153. PMID 34204096
- [Background] Loe H. The Gingival Index, the Plaque Index and the Retention Index Systems. J Periodontol. 1967 Nov-Dec;38(6):Suppl:610-6. doi: 10.1902/jop.1967.38.6.610. No abstract available. PMID 5237684